CLINICAL TRIAL: NCT05164523
Title: The Effect of SGLT2 Inhibitors on Heart Rate Variability, Sympathetic and Parasympathetic Activity and a Neuroinflammatory Biomarker, Brain-Derived Neurotrophic Factor Levels in Patients With Type 2 Diabetes
Brief Title: The Effect of SGLT2 Inhibitors on Heart Rate Variability and BDNF Levels in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Goztepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ayse N Erbakan, Principal Investigator, Goztepe Training and Research Hospital
Other Study IDs: Heart Rate Variability-BDNF
Record Dates: First submitted 2021-10-17; First posted 2021-12-20 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Type 2 Diabetes; Heart Rate Variability
Keywords: type 2 diabetes; SGLT2 inhibitors; heart rate variability; sympathic activity; parasympathetic activity
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with type 2 diabetes treated with SGLT2 inhibitors: metformin using patients with type 2 diabetes who were recently prescribed an SGLT2 inhibitor
  Interventions: Diagnostic Test: 24-hour rhythm Holter; Diagnostic Test: 36 item Short Form Survey (SF-36)
- Patients with type 2 diabetes treated with other oral agents: metformin using patients with type 2 diabetes who were recently prescribed a pre-defined antidiabetic medication other than SGLT2 inhibitors
  Interventions: Diagnostic Test: 24-hour rhythm Holter; Diagnostic Test: 36 item Short Form Survey (SF-36)

INTERVENTIONS:
Diagnostic Test: 24-hour rhythm Holter — Before starting their newly prescribed medication, the investigators will apply 24-hour rhythm Holter and repeat it at the end of the trial.
Diagnostic Test: 36 item Short Form Survey (SF-36) — Before starting their newly prescribed medication, the investigators will apply SF-36 survey and repeat it at the end of the trial.
  Other Names: SF-36

SUMMARY:
Cardiac autonomic neuropathy (CAN) in diabetic patients is an indicator of autonomic nervous system dysfunction and is an important marker for cardiovascular events. Very promising results have been obtained with SGLT2 inhibitors in both cardiac and renal outcomes. The aim is to examine the effects of SGLT2 inhibitor use on cardiac autonomic neuropathy, heart rate variability, sympathetic and parasympathetic nervous system parameters, and their relationship with BDNF levels, one of the neuroinflammatory markers.

DETAILED DESCRIPTION:
Cardiac autonomic neuropathy (CAN) in diabetic patients is an indicator of autonomic nervous system dysfunction and is an important marker for cardiovascular events. Five-year mortality rates of diabetic patients with CAN are significantly higher than those without. Although there are various methods, primarily scintigraphic and pharmacological tests, to evaluate CAN, the practical use of these methods remains limited. In recent years, heart rate recovery (HRR) and heart rate variability (HRV) have been increasingly used as simple, inexpensive, and non-invasive methods to evaluate the status of heart sympathetic and vagus nerve functions. Values obtained as a result of 24-hour rhythm Holter provide the measurement of sympathetic and parasympathetic activity. While a significant relationship was observed between blood glucose levels and HRV in previous studies, no relationship was found between HbA1c levels and HRV.

Brain-derived neurotrophic factor (BDNF) is a member of the neurotrophin family with growth factor properties. Studies with SGLT2 inhibitors have shown a decrease in HbA1c values, weight loss, and a decrease in both systolic and diastolic blood pressure. Very promising results have been obtained with SGLT2 inhibitors in both cardiac and renal outcomes. As a result of these data, these medications are recommended as drugs that should be used in the foreground following metformin, especially in diabetic patients with cardiac and renal diseases. In the study of Shimuz et al. in which the effects of empagliflozin and placebo on heart rate variability were compared in patients with acute myocardial infarction, HRV improved significantly with the use of empagliflozin in the early period. A study examining the effects of empagliflozin use on HRV in patients with type 2 diabetes is still ongoing. Apart from these 2 studies, no study was found in the literature.

The aim of this study is to examine the effects of SGLT2 inhibitor use on cardiac autonomic neuropathy, heart rate variability, sympathetic and parasympathetic nervous system parameters, and their relationship with BDNF levels, one of the neuroinflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* giving consent
* being 30 years old or older
* HbA1c concentrations between 6.5% and 8%
* using metformin as a single agent for at least 3 months
* diabetes age <10 years

Exclusion Criteria: existence of one of the listed conditions:

* having uncontrolled hypothyroidism, hyperthyroidism, or other diseases that may affect cognitive functions
* ketoacidosis or coma
* cerebrovascular disease or psychiatric disorder
* mental retardation, psychosis, dementia, brain trauma, epilepsy and other cerebral diseases
* alcohol or other substance abuse
* hearing loss
* Presence of diseases that will affect cognitive function such as chronic inflammatory diseases and respiratory system diseases
* chronic kidney failure (GFR <45)
* sleep apnea syndrome
* malignancy
* using a sulfonylurea or glinide
* using beta blocker or non-dihydropyridine group calcium antagonists
* diabetic autonomous neuropathy
* atrial fibrillation
* an acute coronary event within the last 3 months

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who refer to a diabetes outpatients clinics to an university hospital
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Heart rate variability parameters | Six months
  The investigators will evaluate the effects of SGLT2 inhibitor use on heart rate variability derived from 24-hour rhythm Holter compared with other antidiabetic medications.
BDNF concentrations | Six months
  The investigators will observe the effects of SGLT2 inhibitors and other oral antidiabetic agents on BDNF levels in type 2 diabetic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse N Erbakan, MD, Principal Investigator — Istanbul Medeniyet University Goztepe Research and TRaining Hospital
Locations (1):
- Istanbul Medeniyet University Goztepe Research and Training Hospital, Istanbul, Turkey (Türkiye)